CLINICAL TRIAL: NCT04079556
Title: Reducing Breast Cancer Risk in Korean American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Korean Community Center of the East Bay (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CBCRP 23AB-1400
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Secondhand Tobacco Smoke Exposure Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tobacco LHW (Experimental): Quit Smoking For a Healthy Family - family-based psycho-education intervention using lay health worker (LHW) outreach.
  Interventions: Behavioral: Tobacco LHW

INTERVENTIONS:
Behavioral: Tobacco LHW — Quit Smoking For a Healthy Family - This is a family-based psycho-education intervention using lay health worker (LHW) outreach. LHW will be trained to recruit smoke-family dyads and provide education and information about tobacco and health, and smoking cessation resources through 2 small-group education sessions and 2 individual phone calls over a 2-month period.

SUMMARY:
The goals of the study are to develop a culturally and linguistically appropriate intervention to reduce SHS exposure for LEP Korean women using a family-focused intervention approach targeting Korean Americans ages 18 and above in the greater San Francisco Bay Area, CA, and to evaluate efficacy of the proposed intervention. The study is a single group feasibility trial targeting a total of 4 lay health workers (LHW) and 24 dyads of LEP Korean women with self-reported SHS exposure at home and a male household smoker. The hypothesis is:

H. Can a family-based intervention approach reduce SHS exposure among Korean American women who live with a current smoker?

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Korean or Korean American;
* Korean speaking;
* reside in the San Francisco Bay Area
* plan to stay in the area for the next 3 months
* for women participants, the participant must report having SHS exposure at home at least 1 day in the past 7 days and live in the same household as the smoker participant to form a dyad.
* for the smoker participants, they must be male and have smoked at least 1 cigarette daily in the past 7 days.
* provide a valid contact telephone number for pre- and post-intervention assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Recruiting for male smokers and female household partner.
Enrollment: 48 (Actual)
Dates: Start 2019-03-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
SHS exposure of non-smokers | 3-month
  biochemically verified 7-day point prevalence of SHS exposure at 3-month post baseline (initiation of intervention)

SECONDARY OUTCOMES:
Smoker's adoption of smoke-free rules | 3-month
  Self-report of adoption of smoke-free home or car rules since program initiation
Smoker's Utilization of smoking cessation resources | 3-month
  Use of evidence-based smoking cessation resources since program initiation
Smoking Abstinence | 3-month
  biochemically verified 7-day point prevalence of SHS exposure at 3-month post baseline (initiation of intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Y Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Korean Community Center of the East Bay, San Leandro, California, United States